CLINICAL TRIAL: NCT04845113
Title: Idiopathic Purpura Fulminans Associated With Anti-PS Antibodies in Children: a French Multicenter Retrospective Study
Brief Title: Idiopathic Purpura Fulminans Associated With Anti-PS Antibodies in Children
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0234
Record Dates: First submitted 2021-04-13; First posted 2021-04-14 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Purpura
Keywords: Protein S acquired deficiency; Idiopathic purpura fulminans
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Acquired Protein S Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Idiopathic purpura fulminans by anti-protein S antibody is a very rare but potentially extremely serious entity. The data in the literature are poor with only isolated report boxes and a single series of less than 10 boxes. The creation of a larger series of cases would make it possible to better understand this pathology and to offer assistance in diagnosis and management.

ELIGIBILITY:
Inclusion criteria:

* diagnostic of idiopathic purpura fulminans
* Acquired protein S deficiency

Exclusion criteria:

- Other infecious purpura diagnosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with diagnostic of idiopathic purpura fulminans and acquired protein S deficiency
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of anti-protein S antibody | 1 day
  Rate of anti-protein S antibody

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre THERON, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC